CLINICAL TRIAL: NCT02652598
Title: A Proof of Concept Open-label Study to Evaluate the Effects of Tolcapone on Cognitive and Behavioral Dysfunction in Patients With Traumatic Brain Injury (TBI), Other Acquired Brain Injuries (ABI), or a Diagnosis of Neurocognitive Disorder (NCD)
Brief Title: Evaluate the Effects of Tolcapone on Cognitive and Behavioral Dysfunction in Patients With BI and NCD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Lieber Institute for Brain Development (LIBD) (Unknown)
Responsible Party: Principal Investigator, Robert Schloesser, MD, Executive Director of Sheppard Pratt-Lieber Research Institute, Inc., Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 805704
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Brain Injuries, Traumatic; Neurocognitive Disorders; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurocognitive Disorders; Brain Injuries | interventions — Tolcapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label (Experimental): Each patient will receive a two-week specified dosing amount of tolcapone (100mg TID on Day 1; 200mg TID on Days 2-14). The patient will be instructed to take the study drug three times daily. Tolcapone will be tapered after Day 14 to avoid potential withdrawal reactions.
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone
  Other Names: Tasmar

SUMMARY:
The experimental design is an open-label two-week trial of tolcapone to evaluate which clinical domains are affected by tolcapone treatment and to identify "responders" to tolcapone treatment in the two subject groups (BI and NCD)

DETAILED DESCRIPTION:
Each patient will receive a two-week specified dosing amount of tolcapone (100mg TID on Day 1; 200mg TID on Days 2-14). The patient will be instructed to take the study drug three times daily. Tolcapone will be tapered after Day 14 to avoid potential withdrawal reactions.

Clinical Instruments for patients:

* Question banks from large patient-reported outcome measure initiatives will be used and administered and used by computerized-adaptive tests (CATs). These include the TBI-QoL for patients with TBI and question banks from the patient-reported outcome measure information systems (PROMIS) and neurology quality of life measurement initiative (Neuro-QoL). Patients will answer questions related to their mobility, fatigue, pain interference, positive affect and well-being, depression, anxiety, anger and irritability, and emotional and behavioral dyscontrol.
* Clinical Global Impressions Scale
* Geriatric Depression Scale-15
* State-Trait Anxiety Inventory
* Hopkins Adult Reading Test
* Frontal Systems Behavior Scale
* Montreal Cognitive Assessment
* Trails A&B
* Modified Wisconsin Card Sorting Test
* NIH Toolbox
* Perceptual Comparison Test
* Brief Test of Attention
* Hopkins Verbal Learning Test
* Brief Visuospatial Memory Test
* Calibrated Ideational Fluency Assessment
* Profile of Mood States
* Digit Span

Clinical Instruments for Informants:

* Neuropsychiatry Inventory
* Apathy evaluation scale
* Overt aggression scale
* Frontal Systems Behavior Scale

Laboratory Measures:

* Blood sample for genotyping
* Blood sample for assessing COMT activity.
* Blood sample for a laboratory profile including CBC, CMP, TSH, Hepatitis Panel (B and C), and RPR
* A urine analysis, urine drug screen, and a urine pregnancy test
* In addition for NCD patients: a blood sample for tests including Serum Calcium, B12, ESR, and C-reactive protein

ELIGIBILITY:
TBI and ABI Patients Inclusion Criteria

* Age 18-70
* Diagnosis of mild, moderate, or severe TBI, or history of ABI with classification to be made based on parameters at the time of the index event or acquired brain injury.
* Index event resulting in Traumatic or Acquired Head Injury occurred >12 months prior to trial initiation
* A current or former patient at the clinics of the Sheppard Pratt Neuropsychiatry Program or another Sheppard Pratt outpatient clinic with medical documentation of TBI or ABI
* Proficient in the English language
* Available to come to Sheppard Pratt Towson for the baseline evaluation and testing and for the duration of the protocol
* Stable neurological and psychiatric symptomatology for 2 months prior to trial initiation as determined by the referring Sheppard Pratt physician.
* Stable medication dose and regimen for 2 months

NCD Patients Inclusion Criteria

* Age 60-75
* NCD diagnosed by a Sheppard Pratt physician, per DSM-5
* No abnormalities on other serum tests to rule out other cause of cognitive impairment: TSH, B12, CBC, Chemistry screen, and RPR.
* Recent structural neuroimaging (within 1 year or since the time of the onset of cognitive complaint)-noncontrast head CT or MRI-to rule out any gross lesion inconsistent with the diagnosis of MCI (e.g. subdural hematoma, normal pressure hydrocephalus, demyelinating lesion, infarct, or mass lesion)
* Proficient in the English language
* A current or former patient at the clinics of the Sheppard Pratt Neuropsychiatry Program or another Sheppard Pratt outpatient clinic with medical documentation of NCD
* Available to come to Sheppard Pratt Towson for the baseline evaluation and testing and for the duration of the protocol
* Stable neurological and psychiatric symptomatology for 2 months prior to trial initiation as determined by the impression of the referring Sheppard Pratt physician.
* Stable medication dose and regimen for 2 months

Exclusion Criteria for All Patients:

* History of, or active, liver disease or abnormal liver function tests--if the patient currently has elevated Alanine Transaminase (ALT) or Aspartate Transaminase (AST) levels that exceed 2 times the upper limit of normal [Normal Reference Ranges ALT (Male: 4-40 IU/L, Female: 4-40 IU/L), AST (Male: 4-31 IU/L, Female: 4-37 IU/L) or the ratio of AST:ALT has exceeded 2:1
* Active alcohol use disorder, as defined by DSM-5, of any severity mild, moderate, or severe
* History of, or active, cardiovascular disease defined as: coronary heart disease, manifested by myocardial infarction, angina pectoris, or heart failure
* Uncontrolled hypo-or hypertension based on Joint National Committee criteria (JNC7) Hypotension: Systolic<90mmHg or diastolic<60mmHg Hypertension: Systolic >140mmHg or diastolic>90 mmHg)
* History of extra-pyramidal symptoms (e.g. tardive dyskinesia, neuroleptic malignant syndrome, or QT prolongation) while on a first-generation anti-psychotic
* Active illicit substance use, resulting in a substance use disorder as defined by DSM-5, of any severity mild, moderate, or severe
* Patient is currently taking tolcapone or any of the following medications that can interact with tolcapone resulting in an adverse events: another COMT inhibitor, benserazide, α-methyldopa, dobutamine, apomorphine, isoproterenol, clozapine, MAO inhibitor
* Known allergy or serious adverse reaction to tolcapone
* Participated in any investigational drug trial in the past 30 days.
* Pregnant or planning to become pregnant during the study period
* Breastfeeding or planning to breastfeed during the study period.

Other Exclusion Criteria for TBI Patients

• Presence of pre-morbid/pre-TBI cognitive impairment or behavioral dysfunction, as per informant or medical documentation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Clinical Global Impression Scale (CGI) to two weeks after medication administration | Up to 2 weeks

SECONDARY OUTCOMES:
Change from Baseline TBI-QoL to two weeks after medication administration | Up to 2 weeks
  Questions from the TBI-QoL battery, which consists of tests to assess items on domains of emotion, social activity, physical activity, and cognition
Change from Baseline NIH Toolbox Cognition Battery to two weeks after medication administration | Up to 2 weeks
  A cognition battery developed by NIH, which consists of tests to assess Executive Function, Attention, Episodic Memory, Language, Processing Speed and Working Memory.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Schloesser, MD, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Baltimore, Maryland, United States